CLINICAL TRIAL: NCT05872204
Title: A Phase II, Open-label, Multicenter Study of Abemaciclib and Letrozole in Patients With Estrogen Receptor-positive Rare Ovarian Cancer
Brief Title: Abemaciclib and Letrozole in Patients With Estrogen Receptor-positive Rare Ovarian Cancer
Acronym: ALEPRO
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Kom Op Tegen Kanker (Other); Eli Lilly and Company (Industry); European Network of Gynaecological Oncological Trial Groups (ENGOT) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S66468
Record Dates: First submitted 2023-05-02; First posted 2023-05-24 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2024-06

CONDITIONS: Low Grade Serous Ovarian Carcinoma; Adult Type Granulosa Cell Tumor
MeSH Terms: interventions — abemaciclib; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Abemaciclib and letrozole (Experimental): Participants received abemaciclib 150 mg tablet orally twice daily and letrozole tablet 2.5 mg orally once daily until disease progression, unacceptable adverse event(s) or death.
  Interventions: Drug: Abemaciclib; Drug: Letrozole

INTERVENTIONS:
Drug: Abemaciclib — 150 mg tablet twice daily
  Other Names: Verzenios
Drug: Letrozole — 2.5 mg tablet once daily
  Other Names: Femara

SUMMARY:
The purpose of this study is to assess the efficacy and safety of abemaciclib and letrozole for treatment of estrogen receptor-positive rare ovarian cancer.

DETAILED DESCRIPTION:
Patients with recurrent, persistent and/or metastatic estrogen receptor-positive rare ovarian cancer, who failed one line of platinum based chemotherapy for advanced or recurrent disease, will be included in this study. One cohort will include low-grade serous or endometrioid epithelial ovarian cancer and another cohort will include adult type granulosa cell tumors. The results of large randomized phase 3 trials of the combination of an aromatase inhibitor combined with a CDK4/6 inhibitor in hormone sensitive, HER2 negative breast cancer can form the basis for a trial with this drug combination in hormone sensitive rare ovarian cancer. The aim is to increase the response rate to aromatase inhibitors and the duration of response in this study population with limited therapeutic options, monitor the quality of life and explore the (epi)genomic signatures that correlate with response or endocrine resistance. Abemaciclib will be supplied as capsules administered orally, 150 mg every 12 hours (Q12H) on Days 1 to 28 of a 28-day cycle, plus letrozole 2.5 mg OD Days 1 to 28 of a 28-day cycle.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary written informed consent of the participant or their legally authorized representative has been obtained prior to any screening procedures.
2. Use of highly effective methods of birth control; defined as those that, alone or in combination, result in low failure rate (i.e., less than 1% per year) when used consistently and correctly; such as implants, injectables, combined oral contraceptives, some IUDs, true sexual abstinence (i.e. refraining from heterosexual intercourse during the entire period of risk associated with the Trial treatment(s)) or commitment to a vasectomised partner.
3. Histological confirmation of diagnosis of low-grade serous (original diagnosis of low-grade serous carcinoma or original diagnosis of serous borderline tumor with subsequent diagnosis of low-grade serous carcinoma )or low-grade endometrioid carcinoma of ovary, fallopian tube or peritoneum or granulosa-cell tumor of the adult type and ER positivity on immunohistochemistry. In order to prevent inclusion of patients with high-grade serous carcinoma, diagnosis of low-grade serous carcinoma will be verified as part of screening review by a gynecologic pathologist. Tissue for confirmation can be from primary tumor or recurrence.
4. For Stage 1: only patients where platinum is still an option are eligible with no limitations in prior chemotherapy regimens and a maximum of 2 prior endocrine therapy regimens. For Stage 2: a further 20 patients where platinum is still an option will be included, with no limitations in prior chemotherapy regimens and a maximum of 2 prior endocrine therapy regimens. Fifteen patients where platinum is not an option are allowed with no limitations in prior chemotherapy regimens and maximum of 2 prior endocrine therapy regimens. Patients cannot have received chemotherapy for platinum resistant or refractory disease.
5. Age > 18 years at time of study entry.
6. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1.
7. Patient must have recurrent, measurable disease by RECIST v1.1. Measurable disease is defined as at least one lesion that can be accurately measured in at least 1 dimension (longest dimension to be recorded). Each lesion must be ≥10 mm when measured by computed tomography (CT), magnetic resonance imaging (MRI), or caliper measurement by clinical exam or must be ≥20 mm when measured by chest x-ray. Lymph nodes must be >15 mm in short axis when measured by CT or MRI.
8. Pre- and post-treatment tissue biopsy and ct-DNA blood sample are mandatory for translational studies. Tissue from an archival tissue sample or fresh tissue obtained from a core or excisional biopsy of a tumor lesion.
9. Patients who were previously treated with letrozole or another aromatase inhibitor are allowed, but capped at 10 patients in each cohort.
10. Patients who received radiotherapy must have completed and fully recovered from the acute effects of radiotherapy. A washout period of at least 14 days is required between end of radiotherapy and randomization.
11. Patients must not have remaining ovarian function. In women who have at least one retained ovary, menopause must be confirmed with laboratory confirmation. Women who have ovarian function are eligible but must be placed on hormonal suppression after a negative serum or urine human chorionic gonadotropin (hCG) test.
12. Abnormal organ function is permitted. However, patients must have:

    1. absolute neutrophil count ≥1500/mL
    2. platelets ≥100.000/mL
    3. hemoglobin ≥9 g/dL
    4. estimated creatinine clearance ≥ 45 ml/min as calculated using the method standard for the institution
    5. total serum bilirubin ≤1.5 X ULN
    6. aspartate aminotransferase (AST/SGOT) and/or alanine aminotransferase (ALT/SGPT) ≤3 X ULN
    7. alkaline phosphatase ≤2.5x ULN (or ≤5.0x ULN if liver or bone metastases)

Exclusion Criteria:

1. For Stage 1: patients where platinum is not an option and platinum refractory patients are not allowed. For Stage 2: patients with platinum refractory disease are not allowed. Patients who received chemotherapy must have recovered (Common Terminology Criteria for Adverse Events [CTCAE] Grade ≤1) from the acute effects of chemotherapy except for residual alopecia or Grade 2 peripheral neuropathy prior to randomization. A washout period of at least 21 days is required between last chemotherapy dose and randomization (provided the patient did not receive radiotherapy).
2. The patient has serious preexisting medical condition(s) that would preclude participation in this study (for example, interstitial lung disease, severe dyspnea at rest or requiring oxygen therapy, severe renal impairment (e.g. estimated creatinine clearance <30 mL/min), history of major surgical resection involving the stomach or small bowel, or preexisting Crohn's disease or ulcerative colitis or a preexisting chronic condition resulting in baseline Grade 2 or higher diarrhea).
3. Current use of food or drugs known to be potent CYP3A4 inhibitors, drugs known to be potent CYP3A4 inducers (for examples, see the Prohibited Concomitant Medications section).
4. Diagnosis of another malignancy within 3 years, except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ of the cervix.
5. Patient cannot have previously received a prior cyclin dependent kinase inhibitor (CDKi).
6. Known Hepatitis B, Hepatitis C or human immunodeficiency virus (HIV) infection.
7. Inability or unwillingness to swallow pills.
8. Patient has had major surgery within 14 days prior to starting study drug or has not recovered from major side effects (tumor biopsy is not considered as major surgery).
9. Active infection requiring intravenous (IV) antibiotics or antifungals, or other uncontrolled recurrent illness requiring hospitalization.
10. History of any of the following: syncope of cardiovascular etiology, ventricular arrhythmia of pathological origin (including, but not limited to, ventricular tachycardia and ventricular fibrillation), sudden cardiac arrest.
11. Prior hematopoietic stem cell or bone marrow transplantation.
12. Known history of brain metastasis(es) that may be considered active (screening imaging of brain is not required unless there is clinical suspicion of brain metastases). Patients with previously treated brain metastases may participate provided that the lesions are stable (without evidence of progression for at least 12 weeks on imaging), there is no evidence of new or enlarging brain metastases.
13. Known abnormalities in coagulation such as bleeding diathesis, or treatment with anticoagulants precluding intramuscular injections of goserelin (if applicable).
14. Known or possible hypersensitivity to letrozole or abemaciclib or any of their excipients.
15. Pre/perimenopausal women with a known hypersensitivity to gnRH (gonadotropin-releasing hormone) agonists.
16. Patients who are pregnant or breastfeeding.
17. Participation in an interventional Trial with an investigational medicinal product (IMP) or device. The patient has received an experimental treatment in a clinical trial within the last 30 days or 5 half-lives, whichever is longer, prior to randomization, or is currently enrolled in any other type of medical research (for example: medical device) judged by the sponsor not to be scientifically or medically compatible with this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-11-30 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
The overall response rate (ORR) of the combination of abemaciclib and letrozole, according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) | Week 24
  RECIST is a standard system to measure how cancer responds to different treatments, including chemotherapy, immunotherapy, and radiation therapy.
The overall response rate (ORR) of the combination of abemaciclib and letrozole, according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) | 3 years
  RECIST is a standard system to measure how cancer responds to different treatments, including chemotherapy, immunotherapy, and radiation therapy.

SECONDARY OUTCOMES:
The duration of response (DOR) of the combination of abemaciclib and letrozole in the intention-to-treat (ITT) population at Week 24 and 3 years. | Week 24 and 3 years
  The DOR is defined as the time from response until disease progression or death in patients who achieve complete or partial response.
The clinical benefit rate (CBR) of the combination of abemaciclib and letrozole. | Week 24 and 3 years
  The CBR is defined as the proportion of patients with a confirmed complete response (CR), partial response (PR) and stable disease (SD) maintained for at least 24 weeks.
The incidence and severity of adverse events, with severity determined according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events Version 5.0 (CTCAE v5.0). | 3 years
  Based on clinically relevant changes from baseline for vital signs and laboratory findings. CTCAE v5.0 uses a range of grades from 1 to 5:
  Grade 1 = mild Grade 2 = moderate Grade 3 = severe Grade 4 = life-threatening Grade 5 = death
Progression-free survival (PFS). | 3 years
  PFS is defined as the time from start of treatment until disease progression/relapse or death from any cause. If the specific event (disease progression/relapse, death, whatever comes first) does not occur, PFS will be censored at the date of last tumor assessment. In case no tumor assessment is available, patients will conservatively be censored at the date of first letrozole + abemaciclib dose.
Overall survival (OS). | 3 years
  OS is defined as the time from start of treatment until death from any cause. Patients who are still alive at the time of OS analysis will be censored at the last date they were known to be alive.
Change from baseline in health-related quality of life using the EQ-5D-5L questionnaire. | Baseline and 3 years
  The EuroQol Five-Dimension Five-Level Questionnaire (EQ-5D-5L) is a self-assessed, health related, quality of life questionnaire. The scale measures quality of life on a 5-component scale including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
Change from baseline in health-related quality of life using the EORTC QLQ-C30 questionnaire. | Baseline and 3 years
  The EORTC Core Quality of Life questionnaire (EORTC QLQ-C30) is designed to measure cancer patients' physical, psychological and social functions. The questionnaire is composed of multi-item scales and single items.

CONTACTS AND LOCATIONS:
Overall Officials: Els Van Nieuwenhuysen, MD PhD, Principal Investigator — UZ Leuven
Locations (12):
- Belgium (3):
  - CHU de Liège, Liège, Liège
  - UZ Gent, Ghent, Oost-Vlaanderen
  - UZ Leuven, Leuven, Vlaams-Brabant
- France (6):
  - Institut De Cancerologie Strasbourg Europe, Strasbourg, Bas-Rhin
  - Institut Bergonie, Bordeaux, Gironde
  - Institut Universitaire Du Cancer Toulouse-Oncopole, Toulouse, Haute-Garonne
  - Institut De Cancerologie De L'Ouest, Saint-Herblain, Loire-Atlantique
  - Centre Leon Berard, Lyon, Métropole de Lyon
  - Groupe Hospitalier Diaconesses Croix Saint Simon, Paris, Île-de-France Region
- Netherlands (3):
  - University Medical Center Groningen, Groningen, Provincie Groningen
  - Erasmus Medical Center Rotterdam, Rotterdam, South Holland
  - University Medical Center Utrecht, Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ottenbourgs T, van Gorp T, Kridelka F, Baert T, Denys H, Selle F, Baas I, Van Rompuy AS, Lambrechts D, Van Nieuwenhuysen E. A phase II, multicenter, open-label study of abemaciclib and letrozole in patients with estrogen receptor-positive rare ovarian cancer: ALEPRO trial. Int J Gynecol Cancer. 2024 Apr 1;34(4):627-630. doi: 10.1136/ijgc-2023-005189. PMID 38453176